CLINICAL TRIAL: NCT03355651
Title: Prospective Study for Assess Efficacy and Tolerability of an Oral Supplement Based on Collagen, HC-15 and Plasmatic Proteins, in the Recovery of ACL After Surgery: a Multicenter, Randomized, Controlled Trial
Brief Title: Efficacy and Tolerability of a Nutritional Supplement, Plactive Progen, in ACL Reconstruction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: OPK-PLA-2015-01
Record Dates: First submitted 2017-11-10; First posted 2017-11-28 (Actual); Last update posted 2017-11-30 (Actual); Status verified 2017-11

CONDITIONS: ACL Reconstruction
Keywords: Anterior Cruciate Ligament Tears; Dietary Supplementations; Plasma Rich Proteins; Collagen; Chondroitin Sulfate; Hyaluronic Acid
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries | interventions — Estrogens, Conjugated (USP)

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: ACL parasagittal cuts were performed in T1 sequences and analyzed by a blinded musculoskeletal radiologist to improve the quality of the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROGEN Group (Active Comparator): PROGEN + Standard Rehabilitation + ACL reconstruction
  Interventions: Dietary Supplement: PROGEN
- Control Group (No Intervention): Standard Rehabilitation + ACL reconstruction

INTERVENTIONS:
Dietary Supplement: PROGEN — Dietary supplement based on plasma proteins, hydrolyzed collagen, a complex of Hyaluronic Acid - Chondroitin Sulfate (HC-15), and vitamin C
  Arms: PROGEN Group

SUMMARY:
This was a prospective, multicenter, randomized, open-label, phase IV trial to compare the efficacy of supplementation with plasma proteins, hydrolyzed collagen (CH), a complex of HA-CS (HC-15), and vitamin C combined with a standard rehabilitation protocol versus the standard rehabilitation protocol only after arthroscopically-assisted functional ACL reconstruction with hamstrings.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 18 and 55 years with partial or complete anterior cruciate ligament (ACL) rupture, diagnosed clinically and by Magnetic Resonance Imaging (MRI), requiring reconstructive surgery.
* Patients with symptoms of acute or subacute ACL rupture (such as inflammation of the knee and pain with leg movement) or chronic ACL tear, including instability of the knee.
* Patients with ACL ruptures without osteochondral lesions requiring additional surgery.
* Patients with a medical history of therapeutic benefit using analgesic agents.

Exclusion Criteria:

* Patients with concomitant osteochondral pathology.
* Patients treated with intra-articular injections of corticosteroids and/or platelet-rich plasma, or with oral glucosamine, CS, HA or CH in the two months prior to surgery.
* Patients with systemic diseases, those treated with antibiotics or other drugs that might alter the healing process, and those who had undergone arthroscopic lavage in the 90 days prior to surgery.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2015-03-09 (Actual); Primary Completion 2017-02-01 (Actual); Study Completion 2017-03-03 (Actual)

PRIMARY OUTCOMES:
Pain improvement | 90 days
  Assessed using a 100-mm Visual Analog Scale (VAS)

SECONDARY OUTCOMES:
Knee function | 90 days
  Assessed using the International Knee Documentation Committee (IKDC) index. The final score was interpreted as a measure of function, with higher scores representing higher levels of function
Analgesic consumption | 90 days
  Analgesic consumption and frequency of analgesic intake during follow-up
Number of rehabilitation sessions required | 90 days
  Number of required rehabilitation sessions at the end of follow-up.
Maduration of the graft | Day 0, day 90
  Assessed by MRI, by a single blind muskuloskeletal radiologist, using a standard procedure based on ACL oblique parasagittal T1 sequences

OTHER OUTCOMES:
Perceived efficacy and tolerability by both patients and physicians | 90 days
  Perceived efficacy and tolerability were rated by both patients and physicians on a 5-point Likert scale, where higher scores indicated better efficacy and tolerability
Safety | 90 days
  Assessed by means of all adverse events (AE) treatment related, reported at the end of follow-up.

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lopez-Vidriero E, Olive-Vilas R, Lopez-Capape D, Varela-Sende L, Lopez-Vidriero R, Til-Perez L. Efficacy and Tolerability of Progen, a Nutritional Supplement Based on Innovative Plasma Proteins, in ACL Reconstruction: A Multicenter Randomized Controlled Trial. Orthop J Sports Med. 2019 Feb 27;7(2):2325967119827237. doi: 10.1177/2325967119827237. eCollection 2019 Feb. PMID 30834280